CLINICAL TRIAL: NCT00847860
Title: Cilostazol Verse Asprin for Vascular Dementia in Poststroke Patients With White
Brief Title: Cilostazol Verse Asprin for Vascular Dementia in Poststroke Patients With White Matter Lesions
Acronym: CAVAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Zhejiang Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Yining Huang, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neurology-2008-VD
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2009-12

CONDITIONS: Vascular Dementia; Stroke
Keywords: cognition
MeSH Terms: conditions — Dementia, Vascular; Stroke | interventions — Cilostazol; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cilostazol
  Interventions: Drug: Cilostazol
- 2 (Active Comparator): Asprin
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 100 mg bid for 12 months
  Arms: 1
Drug: Aspirin — Aspirin 100 mg qd for 12 months
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of PDE-3 inhibitor, cilostazol, in prevention and treatment of vascular dementia, in those with brain white matter lesions and vascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 40 to 80 years
2. After newly ischemic stroke from 3 months to 2 years
3. Brain CT or MRI shows stroke lesions and white matter lesions, ARWMC(Age Related White Matter Change)>=4
4. Moderate or mild cognitive deficits: MMSE 12-26
5. Vascular or mixed dementia: Hachinski ischemic score>4
6. Moderate or mild disability: MRS<=4,NIHSS<20
7. Informed consent

Exclusion Criteria:

1. Definitive diagnosis of dementia prior to the stroke
2. Cerebral hemorrhage in the past
3. Cerebral embolism result from cardiogenic embolus
4. Critically ills: MRS>4,NIHSS>=20
5. Bed-ridden patient who is hardly discovered newly stroke
6. patient with sever cardiac, hepatic or nephric complication
7. dementia caused not by vascular lesions
8. other diseases disturb the cognitive evaluation
9. susceptibility to varieties of allergen
10. abstain from Cilostazol or Asprin
11. antiplatelet treatment, anticoagulation or fibrinolysis are needed because of other diseases
12. rejected to participate by the patient or the family

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-03; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
changes of the scores of MMSE, MOCA,CDR,and Blessed-Roth | one year

SECONDARY OUTCOMES:
stroke recurrence, other vascular ischemic events, bleeding events | one year

CONTACTS AND LOCATIONS:
Overall Officials: Huang Yining, MD PhD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Shanghai Hua Shan Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Kwan J, Hafdi M, Chiang LLW, Myint PK, Wong LS, Quinn TJ. Antithrombotic therapy to prevent cognitive decline in people with small vessel disease on neuroimaging but without dementia. Cochrane Database Syst Rev. 2022 Jul 14;7(7):CD012269. doi: 10.1002/14651858.CD012269.pub2. PMID 35833913